CLINICAL TRIAL: NCT02275585
Title: Portal Vein Thrombosis in Cirrhosis: A Cohort Sudy
Brief Title: Portal Vein Thrombosis in Cirrhosis
Status: Withdrawn | Type: Observational
Why Stopped: other studies with more patients already publicated
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Diana Horta-Sangenis, MD, Corporacion Parc Tauli
Other Study IDs: CSPT2013628
Record Dates: First submitted 2014-10-21; First posted 2014-10-27 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Hepatic Vein Thrombosis; Cirrhosis
Keywords: Portal vein; Thrombosis; Cirrhosis
MeSH Terms: conditions — Budd-Chiari Syndrome; Fibrosis; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cirrhosis: Patients with cirrhosis will be followed looking about the event of portal vein thrombosis
  Interventions: Other: Event of portal vein thrombosis

INTERVENTIONS:
Other: Event of portal vein thrombosis — There is no intervention over patients. They are followed during 3 years to look after any event of portal vein thrombosis

SUMMARY:
This study evaluates the supervivence of cirrhotic patients that develop portal vein thrombosis in comparison to cirrhotic patients that do not develop portal vein thrombosis.

DETAILED DESCRIPTION:
Patients newly diagnosed with portal vein thrombosis by imaging tests, that evaluate the extent and exclude tumoral origin, will be included (informed consent previously signed).

Anticoagulant treatment will be initiated according to clinical guidelines (if there is no contraindication) first with LMWH (low molecular weight heparin) and later with dicoumarin.

An abdominal CT will be performed to evaluate the extent and exclude tumoral origin; a gastroscopy to evaluate portal hypertension (and do prophylaxis if required) and thrombophilia study.

Patients will be followed by imaging and laboratory tests every 6 months; to evaluate the response to the treatment and detect any cirrhosis complication.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis diagnosed by liver biopsy or non-invasive methods/clinical, analytics or ultrasound usual criteria
* Portal vein thrombosis of newly diagnosed (defined as partial or complete obstruction of splenoportal vessels objectified by imaging with/without symptomatology) ≤ 6 months.
* Over 18 years old
* Want to participate (informed consent)

Exclusion Criteria:

* Pregnant or lactating
* Patients with tumoral vein thrombosis or elevated alpha-fetoprotein or high suspicion of underlying neoplastic disease.
* Thrombocytopenia < 25.000 .
* Patients with cavernomatosis or portal vein thrombosis already known.
* Patient refusal to participate
* Patients already treated with anticoagulants for other diseases (atrial fibrillation, pulmonary thrombosis...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Survival of patients with cirrhosis | 12 months

SECONDARY OUTCOMES:
Complications related with cirrhosis | 12 months
  Number of patients with Complications related with cirrhosis including ascites, hepatic encephalopaty, and variceal bleeding
Complications related with anticoagulation treatment | 12 months
  Number of patients with Complications related with anticoagulation treatment including any haemorragic event
Prevalence of thrombophilic disorders in patients with Portal Vein Thrombosis | 12 months
  To know how many patients with Portal Vein Thrombosis have Thrombophilic disorders